CLINICAL TRIAL: NCT04671303
Title: This Study is To Evaluate the Efficacy and Safety of Anlotinib Hydrochloride Capsule Combined With Furmonertinib Mesylate in First-line Treatment of Advanced No-small Cell Lung Cancer
Brief Title: To Evaluate the Efficacy and Safety of Anlotinib Combined With Furmonertinib Mesylate in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuankai Shi, Director, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AFTN-II-01
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib Hydrochloride Capsule Combined with Furmonertinib Mesylate (Experimental): Anlotinib Hydrochloride Capsule: Oral on an empty stomach, once a day, 1 capsule each time, orally for 2 consecutive weeks, stop for 1 week Furmonertinib Mesylate：The dose of Furmonertinib Mesylate is 80 mg once a day, 2 tablets each time, taken orally on an empty stomach before breakfast.
  Take medicine continuously for 3 weeks (21 days) for 1 cycle.
  Interventions: Drug: Anlotinib Hydrochloride Capsule Combined with Furmonertinib Mesylate

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule Combined with Furmonertinib Mesylate — Anlotinib Hydrochloride Capsule: Oral on an empty stomach, once a day, 1 capsule each time, orally for 2 consecutive weeks, stop for 1 week Furmonertinib Mesylate：The dose of Furmonertinib Mesylate is 80 mg once a day, 2 tablets each time, taken orally on an empty stomach before breakfast.
  Take medicine continuously for 3 weeks (21 days) for 1 cycle.

SUMMARY:
This Study is To Evaluate the Efficacy and Safety of Anlotinib Hydrochloride Capsule Combined with Furmonertinib Mesylate in First-line Treatment of Advanced no-squamous and No-small Cell Lung Cancer with Epidermal Growth Factor Receptor Mutation.

DETAILED DESCRIPTION:
This Study is To Evaluate the Efficacy and Safety of Anlotinib Hydrochloride Capsule Combined with Furmonertinib Mesylate in First-line Treatment of Advanced No-squamous and No-small Cell Lung Cancer with Epidermal Growth Factor Receptor Mutation.

This study is a single arm, phase II study, including 18 to 36 subjects; Common Terminology Criteria for Adverse Events 5.0 standard was used to evaluate adverse events of drugs, and Response Evaluation Criteria In Solid Tumors 1.1 was used to evaluated efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced and/or metastatic NSCLC diagnosed histologically and/or cytologically;
2. Age 18 and above; Eastern Cooperative Oncology Group Physical condition: 0~1; The expected survival time is more than 3 months;
3. The previous report confirmed the presence of an EGFR gene exon 19 deletion mutation or exon 21 L858R mutation, and the investigator verified that the report reflects the patient's current genetic status.
4. There is at least one measurable lesion other than brain lesion defined by Response Evaluation Criteria In Solid Tumors 1.1 standard;
5. The main organs are functioning well,Adequate laboratory indicators.
6. Women of childbearing age should agree to use contraceptives during the study period and for a period of six months after the study; Negative serum or urine pregnancy test within 7 days prior to study inclusion, and must be non-lactating; Male patients should agree to use contraception during the study period and for six months after the end of the study period;
7. Patients voluntarily participated in this study, signed informed consent, and had good compliance.

Exclusion Criteria:

1. Prior history of targeted Epidermal Growth Factor Receptor therapy and anti-angiogenic drugs
2. Received chemical or biological drugs after the diagnosis of advanced stage;
3. Subjects had undergone surgery , radiation therapy or other anticancer therapies within 4 weeks prior to the commencement of study treatment; Subjects who have previously received local radiation therapy may be enrolled if the following conditions are met: more than 4 weeks after the end of radiation therapy ;
4. Within 2 weeks before the start of the study, patients were treated with Chinese medicines
5. Imaging shows that the tumor has invaded the periphery of important blood vessels or the investigator has determined that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study.
6. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage ;
7. Brain metastases with symptoms or symptom control time less than 2 weeks;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of drug therapy | up to 4 weeks
  The probability and severity of first cycle adverse events (AE) and serious adverse events (SAE) (based on Common Terminology Criteria for Adverse Events 5.0) and abnormal laboratory test indicators;

SECONDARY OUTCOMES:
The overall efficacy was assessed by the investigators | up to 48 weeks
  Objective response rate (ORR) assessed by the investigators

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai SHI, Doctor, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No